CLINICAL TRIAL: NCT02981849
Title: Validating Adolescent SBIRT Measures
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Conrad N. Hilton Foundation (Other)
Responsible Party: Principal Investigator, Sharon Levy, Associate Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: P00019608
Record Dates: First submitted 2016-03-17; First posted 2016-12-05 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to address the needs for efficient and informative measurement for evaluating adolescent Screening, Brief Intervention, and Referral to Treatment (SBIRT) strategies. The investigators will undertake a longitudinal cohort study to build and validate a substance specific measurement battery that includes patient-centered and intermediary outcomes which can be integrated into a range of healthcare and research settings. The results of this project will enable evaluation of SBIRT trials and clinical efforts by validating a parsimonious set of measurement tools that can be incorporated into electronic health records. The primary goal of the proposed project is to develop a set of brief, valid tools that will allow both researchers and clinicians to collect information that enables evaluating and refining brief interventions.

The main objective is to define and disseminate a set of brief and easy to administer measures that accurately detect 1) substance use frequency, 2) substance-specific patient centered outcomes and 3) intermediate measures of impact of adolescent SBIRT. The specific aim addressed in this project is to develop and administer an assessment battery that includes novel questions assessing substance use to be validated against criterion standard measures both cross-sectionally and longitudinally.

DETAILED DESCRIPTION:
A policy level mandate now exists to deliver screening, brief intervention, and referral to treatment (SBIRT) to all adolescents in primary care. This mandate is spurred by the imperative to reduce the enormous and preventable morbidity and mortality caused by adolescent substance use. Despite this mandate and the opportunity to reach large cohorts of youth early within primary and specialty pediatric care, SBIRT is not routinely delivered nor used in ways that optimize outcomes. The National Institute on Drug Abuse, National Institute on Alcoholism and Alcohol Abuse, the Substance Use and Mental Health Services Administration and the Hilton Foundation have all included adolescent SBIRT in their research, training and service project portfolios. Lacking validated measures that can be used to assess impacts and guide early action, opportunities to glean the most effective strategies and components of brief interventions are hampered despite these considerable investments. This threatens the relevance and sustainability of this work.

To address the needs for efficient and informative measurement for evaluating adolescent Screening, Brief Intervention, and Referral to Treatment (SBIRT) strategies, the investigators will undertake a longitudinal cohort study to build and validate a substance specific measurement battery that includes patient-centered and intermediary outcomes which can be integrated into a range of healthcare and research settings. This is a construct validity study in which the investigators will be interested in seeing whether a brief set of questions will accurately measure substance use when compared to lengthy gold standard measures. This is also a predictive validity study, in which the investigators are interested in seeing whether proposed patient-centered and intermediary outcomes are relevant in predicting future substance use risk or patterns of use. The results of this project will enable evaluation of SBIRT trials and clinical efforts by validating a parsimonious set of measurement tools that can be incorporated into electronic health records.

This project is one component of a two part study in which the investigators will enroll a total of 900 adolescents. The investigators will enroll a total of 450 participants from the Adolescent/Young Adult Medical Clinic for this study and will attempt to follow participant for one year. Accounting for attrition at 6 months and 12 months follow-up, the investigators expect 300 participants will complete the entire study.

ELIGIBILITY:
Inclusion Criteria:

* 14-17 year-old youth presenting for routine medical care at the Adolescent and Young Adult clinic at BCH, with informed assent/consent.
* To be eligible, youth must be between 14-17 years old at the time of enrollment and be able to read and understand English at a middle school level or greater.
* Participants must consent to participation in the study and consent to the 6 month and 12 month follow up assessments.

Exclusion Criteria:

* Patients who are medically or emotionally unstable or otherwise unable to assent/consent at the time of their appointment as determined by their clinician or the research team, those who are unable to speak/read English at a middle school reading level, use a computer keyboard and/or complete an interviewer-assisted questionnaire will be excluded.
* Participants who do not consent to 6 month and 12 month re-assessment will also be excluded.
* Patients who are pregnant at baseline will be excluded from the study.
* If a participant enrolls in the study and becomes pregnant after baseline, the participant will not be excluded from the follow up assessments.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescent, ages 14-17, receiving care at the Adolescent/Young Adult Medicine Clinic at Boston Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2016-01; Primary Completion 2019-03 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Validation of adolescent substance use measures | Past year
  This is a validation project. We aim to validate a single question regarding the frequency of substance against the criterion standard timeline followback calendar
Predictive behaviors that indicate a change in substance use frequency | 1 year
  Change in substance use frequency at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Levy, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No